CLINICAL TRIAL: NCT06369350
Title: Effects of Vitamin B6 on the Exercise Pressor Reflex in Lower Limb Ischemia-Reperfusion
Brief Title: Vitamin B6 on Exercise Pressor Reflex on Leg Ischemia-reperfusion
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Lu Qin, Assistant Professor in Department of Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY000020217; 940567 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2024-04-11; First posted 2024-04-17 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Ischemia Reperfusion Injury; Peripheral Artery Disease
MeSH Terms: conditions — Reperfusion Injury; Peripheral Arterial Disease | interventions — Vitamin B 6

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Vitamin B6 25mg (Active Comparator)
  Interventions: Drug: Vitamin B6 25 MG
- Vitamin B6 50mg (Active Comparator)
  Interventions: Drug: Vitamin B6 50 MG
- Vitamin B6 100mg (Active Comparator)
  Interventions: Drug: Vitamin B6 100 MG

INTERVENTIONS:
Drug: Vitamin B6 25 MG — Vitamin B6 25 mg/day will be given for up to 31 days.
  Arms: Vitamin B6 25mg
Drug: Vitamin B6 50 MG — Vitamin B6 50 mg/day will be given for up to 31 days.
  Arms: Vitamin B6 50mg
Drug: Vitamin B6 100 MG — Vitamin B6 100 mg/day will be given for up to 31 days.
  Arms: Vitamin B6 100mg
Drug: Placebo — Placebo capsule will be given for up to 31 days.
  Arms: Placebo

SUMMARY:
In this study, we are trying to see if vitamin B6 can minimize the amplified blood pressure response to exercise following ischemia-reperfusion injury. We are interested in a protein called P2X3, of which function can be blocked by vitamin B6, in the neurons of our nervous system. It is very important for blood pressure regulation. We would like to see if the P2X3 plays a role in patients' rising blood pressure during exercise. The results of the proposed studies will provide a base for those two potential economic and non-invasive inventions to improve the overall health and well-being of PAD patients.

DETAILED DESCRIPTION:
The Ischemia-reperfusion (IR) injury is caused by a burst of reactive oxygen species (ROS) production during reperfusion, which leads to cell damage and inflammation and further exacerbates the underlying ischemic condition. PAD patients endure this pathological condition during various situations of this disease. In a hindlimb IR model, the blood flow in the lower extremity of the plantar muscle and gastrocnemius muscle reduced at 6 h after the femoral artery ligation and gradually restores at 18, 66 and 114 h after the blood flow reperfusion in the femoral artery. Meanwhile, the mean arterial pressure (MAP) responses to static muscle contraction increased in the above blood reperfusion time courses. Examining the underlying mechanisms leading to the exaggerated EPR in the IR injury of PAD will be essential to provide a fundamental base for developing effective interventions to prevent or alleviate the PAD-associated symptoms and complications. The P2X3 receptor in DRG is a potential candidate for regulating this exaggerated EPR in IR. Vitamin B6 can function as a blockade for the P2 receptors. Therefore, we hypothesize it will attenuate the exaggerated exercise pressor reflex (EPR) in the experimental lower limb IR procedure on healthy human participants.

ELIGIBILITY:
Inclusion Criteria:

* Are males and females at least 21- 70 years of age (inclusive)
* Capable of giving informed consent
* Are of any race or ethnicity
* Can communicate in English
* Females may be on oral contraceptives but will be excluded if they are pregnant or lactating
* Healthy Status as defined by the absence of evidence of any active or chronic disease as determined by the following:
* a detailed medical history
* complete physical examination (including vital signs)
* a blood pressure that is within a safe range (<150/100mmHg)

Exclusion Criteria:

* < 21 years of age or > 70 years of age
* Pregnant or nursing woman
* Prisoners or institutionalized individuals unable to consent
* Decisional impairment
* Not able to communicate in English.
* Current smoker
* Have any clinically relevant history or the presence of metabolic (e.g., diabetes), respiratory, renal, hepatic, gastrointestinal, hematological, lymphatic, neurological, cardiovascular, or other disease or diseases that, in the opinion of the research team, exclude the subject from participation.
* Presenting with a resting blood pressure of 150/100 or higher
* Taking any medications that affect vascular control or autonomic function (e.g. beta blockers, ACE inhibitors, calcium channel blockers, etc.)
* Taking a multivitamin with B6, a B-complex vitamin, or vitamin B-6 at baseline, with a history of Parkinson's disease, and taking levodopa
* Known allergy or hypersensitivity to Vitamin B6
* Opioid Use Disorder or on opioid therapy
* Subject has a recent drug or alcohol abuse history (less than 6 months) or is currently using or abusing excessive alcohol or drugs. Excessive alcohol will be defined as greater than 14 drinks per week. Use of recreational drugs in the past 6 months is also an exclusion.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
baseline blood pressure in mmHg | Recorded continuously for up to 4 hours during the study visit
Second visit blood pressure in mmHg | Recorded continuously for up to 4 hours during the second study visit (up to 31 day after the first visit))
baseline heart Rate in beats per minute | Recorded continuously for up to 4 hours during the study visit
Second visit heart Rate in beats per minute | Recorded continuously for up to 4 hours during the second study visit (up to 31 day after the first visit))
baseline muscle sympathetic nerve activity in burst/min | Recorded continuously for up to 4 hours during the study visit
Second visit muscle sympathetic nerve activity in burst/min | Recorded continuously for up to 4 hours during the second study visit (up to 31 day after the first visit))
baseline walking time in minutes | Recording walking time to fatigue (up to 22 minutes maximum) during the study visit
Second visit walking time in minutes | Recording walking time to fatigue (up to 22 minutes maximum) during the second visit (up to 31 days after the first visit))

CONTACTS AND LOCATIONS:
Overall Officials: Lu Qin, Principal Investigator — Penn State College of Medicine